CLINICAL TRIAL: NCT03677271
Title: Personalised Home-based Physical Activity Intervention in Older Adults With Heart Failure: Advancing Towards an Effective Clinical Therapy
Brief Title: A Novel Home-based Physical Activity Intervention for Stable Chronic Heart Failure Patients
Acronym: PAHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 7512; IRAS project ID: 173307 (Other: NUTH)
Record Dates: First submitted 2018-09-05; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity (Other)
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity

SUMMARY:
The project focuses on heart failure (HF), a complex clinical syndrome of symptoms and signs that suggest the efficiency of the heart as a pump is impaired. Around 950,000 people in the UK have HF. Both the incidence and prevalence of heart failure increase steeply as a result of an ageing population, improved survival of people with ischaemic heart disease and more effective treatments for heart failure. Aside from the obvious individual burden HF also accounts for 1 million inpatient bed days - 2% of all NHS inpatient bed days and 5% of all emergency medical admissions to hospital which are projected to rise by 50% over the next 25 years. There is a pressing need to explore effective ways to manage the individual and societal burden of HF.

Despite exercise being an effective, safe, and a recommended (class I) therapy for people with heart failure according to clinical guidelines from the UK, EU, and USA, it is currently out of reach for majority people with HF. This project addresses this directly by designing and evaluating an exercise therapy that will be available to those living with HF with potential to improve their symptoms, function and quality of life

DETAILED DESCRIPTION:
The present project aligns with Ageing Body Theme of the Newcastle NIHR Biomedical Research Centre. In particular the Chronic Cardiac Disease theme because it focuses on Heart Failure and how to improve clinical care and outcomes, physical function and quality of life of those living with heart failure. The project will develop and evaluate a novel non-pharmacological therapeutic approach (home-based exercise programme with behavioural support) which recognises the complexity of heart failure and the need to treat each individual patient in an optimal way. Such therapy will be tailored for people with heart failure who are, under current clinical care, lacking the well-recognised benefits associated with exercise therapy. After initial evaluation, it is expected that this project will inform development of a large definitive trial (subject to separate funding application) which findings will be translated into clinical care to improve outcomes in people with heart failure. Results of such a trial are expected to have a significant impact on current clinical practice and the development of new cardiac rehabilitation guidelines for heart failure.

It is important to indicate that home-based exercise cardiac rehabilitation programmes have been introduced in an attempt to widen access and participation as an alternative to supervised centre-based rehabilitation in conditions other than heart failure. Home-based exercise programmes are reported to be equally effective as centre based programmes in people with coronary artery disease i.e. following myocardial infarction and/or revascularisation, but remain to be designed and evaluated in those living with heart failure and this is subject to the present investigation

ELIGIBILITY:
Inclusion Criteria:

1. Adults (>50 years of age) with chronic HF due to reduced ejection fraction
2. Clinically stable for at least 6 weeks prior to screening
3. Receipt of optimal medical treatment
4. Able to walk and perform activities of daily living independently
5. New York Heart Association functional class II-IV
6. Left ventricular ejection fraction <40%
7. Willingness to undertake a physical activity intervention
8. Willingness to visit the clinical research facility on 2 separate occasions

Exclusion Criteria:

1. Severe aortic stenosis
2. Severe cardiac arrhythmias
3. Myocardial infarction, percutaneous coronary intervention and/or bypass graft surgery over the past 3 months
4. Severely obese i.e. body mass index >40
5. Implanted with left ventricular assist device
6. Current participation in cardiac rehabilitation programme
7. Inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with heart failure screened, recruited into and completing the intervention | 2 years
  Data will be collected on recruitment and retention rates and adherence to intervention and trial procedures. Collated data will be expressed in percentages.

SECONDARY OUTCOMES:
Quality of Life Score using Minnesota living with heart failure questionnaire | 2 years
  This is a qualitative marker which will be assessed using the Minnesota Living with Heart Failure Questionnaire. Pre and post intervention scores will be analysed to assess differences in this outcome.
Maximum Oxygen Consumption (ml/Kg/min) Post intervention | 2 years
  This is a marker of overall fitness levels and the investigators shall sample data pre and post intervention to assess changes in fitness during the intervention
Haemodynamic markers (cardiac output, stroke Volume) | 2 years
  Cardiac output (L/min) is the amount of blood pumped out of the ventricles per minute while stroke volume (ml/beat) is the amount of blood pumped out of the heart per beat. Both markers gives an indication of cardiac function and higher values during exercise indicates better functioning of the heart. The investigators shall evaluate these markers pre and post intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okwose NC, O'Brien N, Charman S, Cassidy S, Brodie D, Bailey K, MacGowan GA, Jakovljevic DG, Avery L. Overcoming barriers to engagement and adherence to a home-based physical activity intervention for patients with heart failure: a qualitative focus group study. BMJ Open. 2020 Sep 21;10(9):e036382. doi: 10.1136/bmjopen-2019-036382. PMID 32958484

DOCUMENTS (2):
  • Informed Consent Form (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT03677271/ICF_000.pdf
  • Study Protocol (2015-04-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT03677271/Prot_001.pdf